CLINICAL TRIAL: NCT06048991
Title: Evaluation of Thermographic Images of the Knee in Patients With Anterior Cruciate Ligament Reconstruction Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Thermo-LCA
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: ACL Injury
Keywords: ACL reconstruction; Anterior cruciate ligament; infrared thermography; joint inflammation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Knees termographic evaluation (Experimental): All 30 patients will undergo thermographic evaluation of the operated knee of ACL reconstruction and of the controlateral knee.
  Interventions: Diagnostic Test: Thermographic assessment

INTERVENTIONS:
Diagnostic Test: Thermographic assessment — Patients will undergo a termographic evaluation of the operated knee of ACL reconstruction and of the controlateral knee.

SUMMARY:
The Thermo-LCA study is a diagnostic interventional study for assessment of knee temperature of asymptomatic patients with ACL reconstruction compared with unoperated healthy contralateral knee. The aim of the study is to analyze thermographic images obtained from the knees of asymptomatic patients with ACL reconstruction that occurred between the previous 2 and 5 years, to assess the presence of inflammation in the knee with reconstructed ACL compared with the contralateral.

DETAILED DESCRIPTION:
Thermo-LCA study involves recruitment of thirty volunteers with unilateral ACL reconstruction Will be enrolled subjects aged 18 to 40 years, with no history of previous surgery or chronic gonalgia in the contralateral knee. Once the patient's Informed Consent has been obtained, the patient will wait sitting 10 minutes inside the temperature-controlled room of 23°C, a thermographic assessment will then be performed using a FLIRT1020 thermal imaging camera. Photographs will be acquired in anteroposterior, right lateral, left lateral, and posteroanterior views of both knees. The patient will then perform a knee flexion-extension exercise against resistance for 2 minutes using a 2 kg weighted ankle monitor. The speed at which this exercise is performed will be constant for all subjects, with one repetition per second per leg. Following this exercise, four more thermographic images identical to the first will be acquired. Basal thermographic assessments will be performed at 5', 10' and 20' minutes after the end of the exercise.Once the images are acquired these will be analyzed using ResearchIR software, regions of interest of the knees will then be constructed and their temperature change over the various acquisitions and how it changes after physical exertion will then be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged between 18 and 40 years;
2. Asymptomatic at the time of evaluation (IKDC ≥95);
3. No history of previous surgery or contralateral knee fractures;
4. No history of direct or indirect trauma in the previous six months to either knee;
5. Absence of gonalgia (VAS pain equal to 0) at evaluation;
6. BMI between 18.5 kg/m2 and 29.9 kg/m2.

Exclusion Criteria:

1. Patients who are incapacitated or have neurological disorders that may invalidate the research protocol;
2. Diagnosis of leukemia, known presence of metastatic malignant cells, current or planned chemotherapy;
3. Diagnosis of rheumatoid arthritis, Reiter's syndrome, psoriatic arthritis, gout, ankylosing spondylitis or arthritis resulting from another inflammatory disease; human immunodeficiency virus (HIV) infection, viral hepatitis; chondrocalcinosis;
4. Patients with uncontrolled diabetes mellitus;
5. Patients with uncontrolled thyroid metabolic disorders;
6. Patients abusing alcoholic beverages, drugs, or medications;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Total knee temperature | baseline
  By thermographic analysis, the average skin temperature of the entire knee will be assessed, as well as the minimum temperature and maximum temperature.
Temperature of the knee regions of interest | baseline
  The mean skin temperature will be assessed, as well as the minimum and maximum temperature of the regions of interest in the knee, divided into medial, lateral, patellar and supra patellar areas.
The Tegner Activity Level Scale | baseline
  The Tegner Activity Level Scale: allows the estimation of a subject's motor activity level with a score between 0 and 10, where 0 represents 'inability' and 10 represents 'participation in competitive sports, such as soccer at the national or international level. This score is the one most commonly used to define the motor activity level of patients with knee disorders.
IKDC-Subjective Score (Subjective International Knee Documentation Committee) | baseline
  The IKDC-Subjective Score (Subjective International Knee Documentation Committee) is a subjective, knee-specific rating scale.The questionnaire examines 3 categories: symptoms, sports activity, and knee function. The response "Unable to perform any of the above activities due to knee pain" receives a score of 0 while the response "Very strenuous activities like jumping or pivoting as in basketball or soccer" receives a score of 4. This is how item 1, which is related to the highest level of activity without significant pain, is scored. For item 2, which asks about the frequency of pain in the last four weeks, the responses "Constant" and "Never" receive scores of 0 and 10, respectively.
  The IKDC Subjective Knee Evaluation Form is graded by adding the results of each item's scores, and then converting the result to a scale from 0 to 100.If there is a score of 100, it means that there is no restrictions on the daily activities or athletic endeavors and doesn't experience any symptoms.
Objective parameters - Circumferences | baseline
  Bilateral trans- and supra- patellar circumferences measurement for comparative analysis.The measurement will be taken by the orthopedist by meter and will be reported in centimeters
Objective parameters- Range of Motion | baseline
  Evaluation of the Range of Motion for comparative analysis. Range of motion (ROM) is a term used to describe how far you can move a joint or muscle in various directions. It is used to measure how much you can move a joint on your own (active ROM) or with the assistance of someone else (passive ROM).Range of motion is measured using a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Di Martino, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Moses B, Orchard J, Orchard J. Systematic review: Annual incidence of ACL injury and surgery in various populations. Res Sports Med. 2012 Jul;20(3-4):157-79. doi: 10.1080/15438627.2012.680633. PMID 22742074
- [Background] Sanders TL, Maradit Kremers H, Bryan AJ, Larson DR, Dahm DL, Levy BA, Stuart MJ, Krych AJ. Incidence of Anterior Cruciate Ligament Tears and Reconstruction: A 21-Year Population-Based Study. Am J Sports Med. 2016 Jun;44(6):1502-7. doi: 10.1177/0363546516629944. Epub 2016 Feb 26. PMID 26920430
- [Background] Mall NA, Chalmers PN, Moric M, Tanaka MJ, Cole BJ, Bach BR Jr, Paletta GA Jr. Incidence and trends of anterior cruciate ligament reconstruction in the United States. Am J Sports Med. 2014 Oct;42(10):2363-70. doi: 10.1177/0363546514542796. Epub 2014 Aug 1. PMID 25086064
- [Background] Lie MM, Risberg MA, Storheim K, Engebretsen L, Oiestad BE. What's the rate of knee osteoarthritis 10 years after anterior cruciate ligament injury? An updated systematic review. Br J Sports Med. 2019 Sep;53(18):1162-1167. doi: 10.1136/bjsports-2018-099751. Epub 2019 Apr 1. PMID 30936063
- [Background] Ajuied A, Wong F, Smith C, Norris M, Earnshaw P, Back D, Davies A. Anterior cruciate ligament injury and radiologic progression of knee osteoarthritis: a systematic review and meta-analysis. Am J Sports Med. 2014 Sep;42(9):2242-52. doi: 10.1177/0363546513508376. Epub 2013 Nov 8. PMID 24214929
- [Background] Larsson S, Struglics A, Lohmander LS, Frobell R. Surgical reconstruction of ruptured anterior cruciate ligament prolongs trauma-induced increase of inflammatory cytokines in synovial fluid: an exploratory analysis in the KANON trial. Osteoarthritis Cartilage. 2017 Sep;25(9):1443-1451. doi: 10.1016/j.joca.2017.05.009. Epub 2017 May 15. PMID 28522220
- [Background] Roemer FW, Englund M, Turkiewicz A, Struglics A, Guermazi A, Lohmander LS, Larsson S, Frobell R. Molecular and Structural Biomarkers of Inflammation at Two Years After Acute Anterior Cruciate Ligament Injury Do Not Predict Structural Knee Osteoarthritis at Five Years. Arthritis Rheumatol. 2019 Feb;71(2):238-243. doi: 10.1002/art.40687. Epub 2018 Dec 4. PMID 30079991
- [Background] Romano CL, Logoluso N, Dell'Oro F, Elia A, Drago L. Telethermographic findings after uncomplicated and septic total knee replacement. Knee. 2012 Jun;19(3):193-7. doi: 10.1016/j.knee.2011.02.012. Epub 2011 Mar 26. PMID 21441031
- [Background] Ramirez-GarciaLuna JL, Bartlett R, Arriaga-Caballero JE, Fraser RDJ, Saiko G. Infrared Thermography in Wound Care, Surgery, and Sports Medicine: A Review. Front Physiol. 2022 Mar 3;13:838528. doi: 10.3389/fphys.2022.838528. eCollection 2022. PMID 35309080
- [Background] Dias de Lacerda AP, Rodrigues de Andrade P, Kamonseki DH, Parizotto NA, Alves da Silva AS, Bernardo de Medeiros L, de Almeida Ferreira JJ. Accuracy of infrared thermography in detecting tendinopathy: A systematic review with meta-analysis. Phys Ther Sport. 2022 Nov;58:117-125. doi: 10.1016/j.ptsp.2022.10.005. Epub 2022 Oct 10. PMID 36274313
- [Background] Tan YK, Hong C, Li H, Allen JC Jr, Thumboo J. Thermography in rheumatoid arthritis: a comparison with ultrasonography and clinical joint assessment. Clin Radiol. 2020 Dec;75(12):963.e17-963.e22. doi: 10.1016/j.crad.2020.08.017. Epub 2020 Sep 13. PMID 32938539
- [Background] Umapathy S, Thulasi R, Gupta N, Sivanadhan S. Thermography and colour Doppler ultrasound: a potential complementary diagnostic tool in evaluation of rheumatoid arthritis in the knee region. Biomed Tech (Berl). 2020 May 26;65(3):289-299. doi: 10.1515/bmt-2019-0051. PMID 31821162
- [Background] Denoble AE, Hall N, Pieper CF, Kraus VB. Patellar skin surface temperature by thermography reflects knee osteoarthritis severity. Clin Med Insights Arthritis Musculoskelet Disord. 2010 Oct 15;3:69-75. doi: 10.4137/CMAMD.S5916. PMID 21151853